CLINICAL TRIAL: NCT05317871
Title: Cerebral Clearance Mechanisms in Atypical Neurodegenerative Diseases: A Multi-modal Study on Lymphatic, Glymphatic and Blood-brain-barrier Function
Brief Title: Clearance Mechanisms in Atypical Neurodegenerative Diseases
Acronym: PeptiClear
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Robert Perneczky, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: 21-0106
Record Dates: First submitted 2021-11-02; First posted 2022-04-08 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Neurodegenerative Diseases; Frontotemporal Degeneration
Keywords: Neurodegenerative diseases; Frontotemporal Degeneration; Clearance; Blood-brain-barrier; Sleep; Microglial activation; Glymphatic system
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — APOE-genotyping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lewy Body Spectrum Diseases
- Progressive Supranuclear Palsy
- Corticobasal Syndrome
- Frontotemporal Degeneration

SUMMARY:
The project PeptiClear aims to investigate whether the blood-brain-barrier (BBB) and the glymphatic system are compromised in atypical neurodegenerative diseases, and whether Alzheimer´s disease (AD)-related copathology, vascular lesions or sleep disturbances modify the clinical picture or structural and/or functional features of the diseases.

DETAILED DESCRIPTION:
It is well established for the frequent sporadic (non-genetic) variant of Alzheimer´s disease (AD) that not the overproduction of a specific protein (Amyloid-beta - Aβ) is a major cause but rather the insufficient clearance of this protein from the central nervous system. On one hand, under physiological conditions, the interplay of the several cell types (cerebral endothelial cells, perivascular mural cells (pericytes), glial cells (astrocytes and microglia) and neurons) regulates the neuronal and glial cell environment and is crucial for cell function and survival. On the other hand, Aβ aggregates lead to BBB damage and activation of microglial cells. The BBB facilitates the clearance of proteins such as Aβ via the cerebrovascular system, but its association with other intracerebral Aβ drainage systems, such as the glympathic system, remains to be clarified. As the glymphatic system is mainly active during sleep, sleep disturbances could influence the clinical course. Concerning atypical neurodegenerative diseases, it is not clear whether tau or alpha-synuclein (alpha-syn) deposits also have a potential to damage the BBB. In AD Aβ aggregation and vascular changes give rise to insufficient protein clearance and thus contribute to AD pathogenesis in a synergistic fashion. However the role of copathology in atypical neurodegenerative diseases - which mainly consists of Alzheimer-related changes and vascular pathology - is elusive and remains to be clarified.

The prospective study cohort (N ~80) will include patients with Lewy Body spectrum disease, progressive supranuclear palsy, corticobasal syndrome and frontotemporal dementia. All study participants will undergo a detailed clinical and neuropsychological assessment according to a standardised protocol (i.a. magnet resonance imaging (MRI), positron emission tomography (PET), cerebrospinal fluid (CSF), actigraphy).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Atypical Parkinsonian Disorders or Frontotemporal Dementia
* Able to provide written informed consent
* Unchanged pharmacotherapy within 4 days prior to the study specific assessments
* Fluent in German

Exclusion Criteria:

* Unable to give informed consent or has a legal guardian
* Other severe mental disorder, e.g. schizophrenia or bipolar affective disorder
* Clinically relevant depression
* Acute suicidality
* Current alcohol, drug or medication abuse
* History of severe traumatic brain injury within 3 months prior to inclusion
* Structural lesions of the basal ganglia or brain stem
* Severe neurological disorder including (but not limited to) epilepsy, systemic disorders, stroke, repeated transient ischaemic attacks, increased brain intracranial pressure, normal pressure hydrocephalus
* Severe medical disorders including (but not limited to) heart failure, respiratory failure, uncontrolled severe arterial hypertension
* Electronic implants (e.g. cardiac pacemaker) or other MRI contraindication
* Renal failure > stage 3 (GFR < 30 mL/min)
* Pregnancy
* Unresolved malignancies within two years prior to inclusion
* Severe current infections or other chronic or systemic disorders
* Other circumstances which preclude participation based on the investigator's judgement

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atypical neurodegerative diseases: Lewy-Body Spectrum Diseases, Progressive Supranuclear Palsy, Corticobasal Syndrome, Frontemporal Degeneration
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Disruption of the brain-blood-barrier between the subgroups | Baseline
  Name of Measurement: Ktrans; Measurement Tool: dynamic contrast imaging(DCI) sequence (MRI); Unit: min -1
Clearance mechanisms and glymphatic or cerebral lymphatic system | Baseline
  Name of Measurement: Diffusion tensor imaging (DTI) Analysis along the perivascular space (ALPS); Measurement Tool: DTI MRI; Unit: mean (Dxpro, Dypro)/ mean (Dypro, Dzasc)
Changes in circadian rhythms | Baseline
  Sleep Efficiency, proportional integration mode (PIM) ;Measurement Tool: Actigraphy; Units: counts
Correlation between clinical symptoms, tau pathology and BBB disorder | Baseline
  Correlations between neuropsychological tests (e.g. Clinical Dementia Rating Sum of Boxes), CSF markers (pg/ml) and TAU PET, standardized uptake value ratio (SUVr) and Ktrans map

CONTACTS AND LOCATIONS:
Overall Officials: Robert Perneczky, Prof. Dr., Principal Investigator — Klinik und Poliklinik für Psychiatrie und Psychotherapie des LMU Klinikums
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie des LMU Klinikums, München, Bavaria, Germany